CLINICAL TRIAL: NCT03327584
Title: Ultrasound Guided Versus Landmark Guided Small & Medium Joint Arthrocentesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24623
Record Dates: First submitted 2017-10-27; First posted 2017-10-31 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Effusion Joint
MeSH Terms: conditions — Hydrarthrosis | interventions — Arthrocentesis

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound Guided Arthrocentesis (Active Comparator): The patients in this group will have ultrasound guided arthrocentesis.
  Interventions: Procedure: Arthrocentesis
- Landmark Guided Arthrocentesis (Active Comparator): The patients in this group will have landmark guided arthrocentesis.
  Interventions: Procedure: Arthrocentesis

INTERVENTIONS:
Procedure: Arthrocentesis — Athrocentesis

SUMMARY:
Arthrocentesis is the removal of synovial fluid for analysis of pathologic processes. Small & medium joint arthrocentesis will be defined as the following joints: elbow, wrist, finger, ankle and toe. Ultrasound (US) and landmark (LM) small & medium joint arthrocentesis are both performed within the clinical setting. Both techniques are considered standard of care. Selection of which technique to use is dependent upon the physician's preference. There is currently limited data comparing the two methods. The investigators hope to determine if one modality is more effective in terms of success rate, number of attempts, and time to complete the procedure.

DETAILED DESCRIPTION:
Patients presenting to the Emergency Department who are 18 years old or older, who do not belong to a vulnerable group, requiring small or medium joint arthrocentesis will be included in this trial. The investigators will randomize each patient into LM vs US. Data collected will include number of attempts to tap the joint, success rate, and time for procedure to be completed. The arthrocentesis will be performed by PGY-3 residents only. A 21 gauge needle will be used for the arthrocentesis.

ELIGIBILITY:
Inclusion Criteria:

* All patients who require an arthrocentesis of a small and/or medium joint (defined previously)

Exclusion Criteria:

* Coagulopathic patients
* Patients on anticoagulants
* Patients with cellulitis overlying the joint.
* Patients with artificial joints
* Adults Unable to Consent
* Vulnerable Populations

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Superiority of Method of arthrocentesis | 1 day
  Number of attempts until successful arthrocentesis

SECONDARY OUTCOMES:
Success of method | 1 day
  Completion of arthrocentesis after three attempts

CONTACTS AND LOCATIONS:
Overall Officials: Ryan C Gibbons, MD, Principal Investigator — Lewis Katz School of Medicine at Temple University
Locations (1):
- Lewis Katz School of Medicine at Temple University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gibbons RC, Zanaboni A, Genninger J, Costantino TG. Ultrasound-versus landmark-guided medium-sized joint arthrocentesis: A randomized clinical trial. Acad Emerg Med. 2022 Feb;29(2):159-163. doi: 10.1111/acem.14396. Epub 2021 Oct 23. PMID 34608713